CLINICAL TRIAL: NCT00557362
Title: Mycotic Ulcer Treatment Trial Therapeutic Exploratory Study
Brief Title: Therapeutic Exploratory Study of Comparing Natamycin and Voriconazole to Treat Fungal Corneal Ulcer
Acronym: MUTT_TE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: That Man May See, Inc. (Other); Aravind Eye Hospitals, India (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H9332-31301-01
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Fungal Keratitis
Keywords: Keratitis; Eye Infection, Fungal; Fungal Eye Infection; Ocular Infection, Fungal; Fungal Keratitis; Mycotic Infections, Ocular; Voriconazole; Natamycin
MeSH Terms: conditions — Keratitis; Eye Infections, Fungal | interventions — Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Topical voriconazole with corneal de-epithelialization
  Interventions: Drug: Voriconazole; Procedure: Corneal de-epithelialization
- 2 (Active Comparator): Topical voriconazole without corneal de-epithelialization
  Interventions: Drug: Voriconazole
- 3 (Active Comparator): Topical natamycin with corneal de-epithelialization
  Interventions: Drug: Natamycin 5%; Procedure: Corneal de-epithelialization
- 4 (Active Comparator): Topical natamycin without corneal de-epithelialization
  Interventions: Drug: Natamycin 5%

INTERVENTIONS:
Drug: Natamycin 5% — One drop of medication will be given every one hour while awake for one week. For another 2 weeks, one drop of medication should be given every 2 hours while awake
  Arms: 3; 4
Drug: Voriconazole — Voriconazole (VFEND® I.V., Pfizer, New York, NY) will be prepared as a 1% solution.
  One drop of medication should be given every one hour while awake for one week. For another 2 weeks, one drop of medication should be given every 2 hours while awake
  Arms: 1; 2
Procedure: Corneal de-epithelialization — Corneal de-epithelialization at 1 week and 2 weeks from enrollment to increase epithelial penetration of antifungal medications.
  Arms: 1; 3

SUMMARY:
We evaluated whether voriconazole is a superior treatment to natamycin for filamentous fungal keratitis in a randomized, masked, controlled trial. This is a therapeutic exploratory study to investigate the safety and feasibility of conducting a larger study and to generate preliminary data.

DETAILED DESCRIPTION:
Fungal ulcers tend to have very poor outcomes with the most common treatments, amphotericin B and natamycin. There has been only a single randomized trial of anti-fungal therapy for fungal ulcers and no new medications have been approved by the FDA since the 1960s. There are studies that indicate that the newer triazoles, such as voriconazole, are more effective in vitro against filamentous fungi such as Aspergillus spp., a common cause of fungal keratitis1-3. Despite a number of case reports and in vitro studies, there has been no systematic attempt to determine whether it is more or less effective clinically than natamycin, the only commercially available FDA-approved agent. There is little data available for physicians to make an informed, evidence-based decision on choice of antifungal.

We evaluated whether voriconazole is a superior treatment to natamycin for filamentous fungal keratitis in a randomized, masked, controlled trial. This is a therapeutic exploratory study to investigate the safety and feasibility of conducting a larger study and to generate preliminary data. The primary outcome is visual acuity at 3 months from enrollment. A subset of patients will be followed at 4 years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a corneal ulcer at presentation
* Evidence of filamentous fungus on KOH (or Giemsa or any other stain) or culture
* The patient must be able to verbalize a basic understanding of the study after it is explained to the patient, as determined by physician examiner. This understanding must include a commitment to return for follow-up visits.
* Willingness to be treated as an in-patient or to be treated as an out-patient and come back every 48-72 hours to receive fresh medication for 3 weeks
* Appropriate consent

Exclusion Criteria:

* Overlying epithelial defect < 0.5 mm at its greatest width at presentation
* Impending perforation
* Evidence of bacteria on Gram stain at the time of enrollment
* Evidence of acanthamoeba by stain
* Evidence of herpetic keratitis by history or exam
* Corneal scar not easily distinguishable from current ulcer
* Age less than 16 years (before 16th birthday)
* Bilateral ulcers
* Previous penetrating keratoplasty in the affected eye
* Pregnancy (by history or urine test) or breast-feeding (by history)
* Acuity worse than 6/60 (20/200) in the fellow eye (note that any acuity, uncorrected, corrected, pinhole, or BSCVA 6/60 or better qualifies for enrollment)
* Known allergy to study medications (antifungal or preservative)
* No light perception in the affected eye
* Not willing to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Lietman, MD, Principal Investigator — Proctor Foundation, University of California, San Francisco; Nisha Acharya, MD MS, Principal Investigator — Proctor Foundation, University of California, San Francisco; N V Prajna, MD, Study Director — Aravind Eye Hospital, India
Locations (2):
- India (2):
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Aravind Eye Hospital, Pondicherry, Tamil Nadu

REFERENCES:
- [Derived] Prajna NV, Mascarenhas J, Krishnan T, Reddy PR, Prajna L, Srinivasan M, Vaitilingam CM, Hong KC, Lee SM, McLeod SD, Zegans ME, Porco TC, Lietman TM, Acharya NR. Comparison of natamycin and voriconazole for the treatment of fungal keratitis. Arch Ophthalmol. 2010 Jun;128(6):672-8. doi: 10.1001/archophthalmol.2010.102. PMID 20547942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 27, 2007 to May 12, 2008, all patients with a corneal ulcer presenting to Aravind Eye Hospital's cornea clinics in Madurai and Pondicherry, India, were evaluated for eligibility. The Aravind Eye Care System is both a primary and tertiary care eye hospital in South India with a well-established cornea subspecialty clinic.
Pre-assignment Details: All patients with a corneal ulcer had corneal scrapings using a Kimura spatula for Gram stain and potassium hydroxide wet mount and had cultures plated on blood, chocolate, and potato dextrose agar. If all inclusion criteria and no exclusion criteria were met, the patient was enrolled in the study.
Groups:
- Topical Natamycin With Corneal De-epithelialization: Topical natamycin with corneal de-epithelialization.
  Drug: Natamycin 5% One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
  Procedure/Surgery: Corneal de-epithelialization Corneal de-epithelialization at 1 week and 2 weeks from enrollment to increase epithelial penetration of antifungal medications.
- Topical Natamycin Without Corneal De-epithelialization: Topical natamycin without corneal de-epithelialization.
  Drug: Natamycin 5% One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
- Topical Voriconazole With Corneal De-epithelialization: Topical voriconazole with corneal de-epithelialization.
  Drug: Voriconazole Voriconazole prepared as a 1% solution.
  One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
  Procedure/Surgery: Corneal de-epithelialization Corneal de-epithelialization at 1 week and 2 weeks from enrollment to increase epithelial penetration of antifungal medications.
- Topical Voriconazole Without Corneal De-epithelialization: Topical voriconazole without corneal de-epithelialization.
  Drug: Voriconazole Voriconazole prepared as a 1% solution.
  One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
Period: Overall Study
Arm/Group | Topical Natamycin With Corneal De-epithelialization | Topical Natamycin Without Corneal De-epithelialization | Topical Voriconazole With Corneal De-epithelialization | Topical Voriconazole Without Corneal De-epithelialization
Started | 30 | 30 | 30 | 30
Completed | 28 | 28 | 26 | 27
Not Completed | 2 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Topical Voriconazole With Corneal De-epithelialization: Drug: Voriconazole Voriconazole prepared as a 1% solution. One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake
  Procedure/Surgery: Corneal de-epithelialization Corneal de-epithelialization at 1 week and 2 weeks from enrollment to increase epithelial penetration of antifungal medications.
- Topical Voriconazole Without Corneal De-epithelialization: Drug: Voriconazole Voriconazole prepared as a 1% solution. One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
- Topical Natamycin With Corneal De-epithelialization: Drug: Natamycin 5% One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
  Procedure/Surgery: Corneal de-epithelialization Corneal de-epithelialization at 1 week and 2 weeks from enrollment to increase epithelial penetration of antifungal medications.
- Topical Natamycin Without Corneal De-epithelialization: Drug: Natamycin 5% One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
- Total: Total of all reporting groups
Arm/Group | Topical Voriconazole With Corneal De-epithelialization | Topical Voriconazole Without Corneal De-epithelialization | Topical Natamycin With Corneal De-epithelialization | Topical Natamycin Without Corneal De-epithelialization | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (14.5) | 45.0 (14.5) | 49.8 (11.9) | 45.9 (13.1) | 46.93 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 7 | 11 | 41
  Male | 16 | 21 | 23 | 19 | 79
Region of Enrollment [Number; unit: participants]
  India | 30 | 30 | 30 | 30 | 120
Enrollment logMAR BSCVA [Mean (Standard Deviation); unit: logMAR] — Best spectacle-corrected visual acuity at time of enrollment measured in logMAR
  logMAR | 0.94 (0.66) | 0.96 (0.66) | 0.87 (0.67) | 0.94 (0.61) | 0.93 (0.64)

OUTCOME MEASURES:

1. Primary Outcome: Best Spectacle Corrected Visual Acuity (BSCVA) 3 Months After Enrollment, Adjusting for Enrollment BSCVA in a Multiple Linear Regression Model
Description: The primary efficacy endpoint was BSCVA at 3 months in the study eye, using a linear regression model with 3-month BSCVA measured in logMAR (logarithm of the Minimum Angle of Resolution) as the outcome variable and treatment arm (voriconazole vs natamycin) and enrollment logMAR BSCVA and corneal de-epithelialization (yes or no) as covariates.
Time Frame: 3 months from enrollment
Measure: Mean (95% Confidence Interval); unit: logMAR
Groups:
- Topical Voriconazole: Drug: Voriconazole Voriconazole prepared as a 1% solution.
  One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
- Topical Natamycin: Drug: Natamycin 5%
  One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
Arm/Group | Topical Voriconazole | Topical Natamycin
Number analyzed (Participants) | 60 | 60
logMAR | 0.61 [0.48 to 0.74] | 0.71 [0.57 to 0.84]
Statistical Analysis 1: Comparison: Topical Voriconazole vs Topical Natamycin; Test type: Superiority or Other; p = 0.29, Regression, Linear; Multiple linear regression model adjusted for enrollment BSCVA and corneal de-epithelialization; Mean Difference (Net) = -0.098, 95% CI 2-sided [-0.28 to 0.083]

2. Secondary Outcome: Time to Resolution of Epithelial Defect
Description: Resolution of epithelial defect was defined as the absence of an epithelial defect with administration of fluorescein. The time to re-epithelialization was compared between the voriconazole and natamycin groups using the Cox proportional hazards model, adjusting for baseline epithelial defect size.
Time Frame: 3 months from enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Topical Voriconazole | Topical Natamycin
Number analyzed (Participants) | 60 | 60
days | 13.07 (7.71) | 15.2 (7.03)
Statistical Analysis 1: Comparison: Topical Voriconazole vs Topical Natamycin; Test type: Superiority or Other; p = 0.40, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.76 to 2.02]

3. Secondary Outcome: Size of Infiltrate/Scar Post-treatment Was Analyzed in a Linear Regression Model Using Enrollment Infiltrate/Scar Size as a Covariate.
Description: Size of infiltrate/scar post-treatment was analyzed in a linear regression model using enrollment infiltrate/scar size as a covariate. No differentiation was made between infiltrate and scar when measuring infiltrate/scar size (measured in mm). For analysis, infiltrate/scar size was characterized by the geometric mean of the longest dimension and the longest perpendicular.
Time Frame: 3 months from enrollment
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Topical Voriconazole: Drug: Voriconazole
  Voriconazole prepared as a 1% solution.
  One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
  Note that 9 patients in the voriconazole arm had home visits conducted as their 3 month follow-up visit and scar size was not able to be obtained for these patients so they are not included in these analyses.
- Topical Natamycin: Drug: Natamycin 5%
  One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
  Note that 5 patients in the natamycin arm had home visits conducted as their 3 month follow-up visit and scar size was not able to be obtained for these patients so they are not included in these analyses.
Arm/Group | Topical Voriconazole | Topical Natamycin
Number analyzed (Participants) | 51 | 55
mm | 4.21 [3.93 to 4.49] | 4.08 [3.81 to 4.35]
Statistical Analysis 1: Comparison: Topical Voriconazole vs Topical Natamycin; Test type: Superiority or Other; p = 0.37, Regression, Linear; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.20 to 0.53]

4. Secondary Outcome: Subgroup Analysis - Best Spectacle-corrected Visual Acuity Examined by Voriconazole and Natamycin Treatment Arms in Subgroups of Fungal Ulcers (Fusarium Spp and Aspergillus Spp).
Description: Two subgroup analyses were conducted by causative organism: 1) best spectacle-corrected visual acuity (BSCVA) by treatment arm among Fusarium ulcers; 2) best spectacle-corrected visual acuity (BSCVA) by treatment arm among Aspergillus ulcers.
Time Frame: 3 months from enrollment
Population: This analysis looks at two different subgroups - Fusarium ulcers and Aspergillus ulcers. There were 44 Fusaruim ulcers enrolled in this trial and analyzed here, 23 of which were randomized to voriconazole and 21 to natamycin. There were 19 Aspergillus ulcers analyzed here, 8 of which were randomized to voriconazole and 11 to natamycin.
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Topical Voriconazole | Topical Natamycin
Number analyzed (Participants) | 31 | 32
logMAR
  BSCVA Fusarium ulcers (n=23 vori; n=21 nata) | 0.58 [0.36 to 0.81] | 0.50 [0.27 to 0.74]
  BSCVA Aspergillus ulcers (n=8 vori; n=11 nata) | 0.48 [0.20 to 0.76] | 0.68 [0.44 to 0.92]
Statistical Analysis 1: Comparison: Topical Voriconazole vs Topical Natamycin; Best spectacle-corrected visual acuity (BSCVA) was examined in a linear regression model with enrollment BSCVA and treatment arm as covariates among a subgroup of ulcers caused by Fusarium spp; Test type: Superiority or Other; p = 0.62, Regression, Linear; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.25 to 0.41]
Statistical Analysis 2: Comparison: Topical Voriconazole vs Topical Natamycin; Best spectacle-corrected visual acuity (BSCVA) was evaluated in a linear regression model with enrollment BSCVA and treatment arm as covariates in a subgroup of ulcers caused by Aspergillus spp; Test type: Superiority or Other; p = 0.26, Regression, Linear; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.57 to 0.17]

5. Secondary Outcome: Best Hard Contact Lens-corrected Visual Acuity 3 Months After Enrollment in a Multiple Linear Regression Model With Enrollment Hard Contact Lens-corrected Visual Acuity as a Covariate
Description: Best hard contact lens-corrected visual acuity 3 months after enrollment was evaluated in a multiple linear regression model with enrollment hard contact lens-corrected visual acuity as a covariate. Visual acuity is reported in logMAR (logarithm of the Minimum Angle of Resolution).
Time Frame: 3 months from enrollment
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Topical Voriconazole | Topical Natamycin
Number analyzed (Participants) | 38 | 40
logMAR | 0.39 [0.26 to 0.54] | 0.46 [0.32 to 0.60]
Statistical Analysis 1: Comparison: Topical Voriconazole vs Topical Natamycin; Test type: Superiority or Other; p = 0.53, Regression, Linear; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.26 to 0.14]

ADVERSE EVENTS:
Groups:
- Topical Voriconazole With Corneal De-epithelialization: Drug: Voriconazole Voriconazole prepared as a 1% solution. One drop of medication every one hour while awake for one week. For another 2 weeks, one drop of medication every 2 hours while awake.
  Procedure/Surgery: Corneal de-epithelialization Corneal de-epithelialization at 1 week and 2 weeks from enrollment to increase epithelial penetration of antifungal medications.
Arm/Group | Topical Voriconazole With Corneal De-epithelialization | Topical Voriconazole Without Corneal De-epithelialization | Topical Natamycin With Corneal De-epithelialization | Topical Natamycin Without Corneal De-epithelialization
Serious Adverse Events (participants affected / at risk) | 6/30 | 5/30 | 8/30 | 1/30
Other Adverse Events (participants affected / at risk) | 2/30 | 5/30 | 2/30 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Voriconazole With Corneal De-epithelialization (N=30) | Topical Voriconazole Without Corneal De-epithelialization (N=30) | Topical Natamycin With Corneal De-epithelialization (N=30) | Topical Natamycin Without Corneal De-epithelialization (N=30)
Corneal perforation (Eye disorders) | 5 (5) | 5 (5) | 8 (8) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Voriconazole With Corneal De-epithelialization (N=30) | Topical Voriconazole Without Corneal De-epithelialization (N=30) | Topical Natamycin With Corneal De-epithelialization (N=30) | Topical Natamycin Without Corneal De-epithelialization (N=30)
Local allergic reaction (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increase in hypopyon (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Increase in infiltrate (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
No resolution of epithelial defect by 21 days (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Reepithelialization was defined as an epithelial defect of less than 0.5 mm with administration of fluorescein.
Progressive corneal thinning (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No